CLINICAL TRIAL: NCT06142461
Title: Safety and Immunogenicity of Human Papillomavirus Quadrivalent Vaccine Administered Intradermally and Intramuscularly Via Needle-Free Injection System
Brief Title: Safety and Immunogenicity of HPV Vaccine Administered Intradermally and Intramuscularly Via Needle-Free Injection System
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in landscape of HPV treatment
Sponsor: PharmaJet, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPV-PJ-01; 1R44CA261326-01A1 (NIH)
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Vaccine Reaction
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label vaccination. Serology samples for immunogenicity assessment are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1: Intradermal needle-free injection (Experimental): Fractional dose (2 x 0.1 mL injections) intradermal administration of Gardasil® using PharmaJet Tropis® Needle-Free Injection System.
  Interventions: Drug: Gardasil; Device: PharmaJet Tropis® Needle-Free Injection System
- 2: Intramuscular needle-free injection (Experimental): Full dose (0.5 mL injection) intramuscular administration of Gardasil® using PharmaJet Stratis® Needle-Free Injection System
  Interventions: Drug: Gardasil; Device: PharmaJet Stratis® Needle-Free Injection System
- 3: Needle and syringe (Active Comparator): Full dose (0.5 mL injection) intramuscular administration of Gardasil® using needle and syringe
  Interventions: Drug: Gardasil

INTERVENTIONS:
Drug: Gardasil — Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant Pre-filled syringe, 0.5mL dose volume
  Other Names: Gardasil PFS, 0.5mL
  Arms: 3: Needle and syringe
Drug: Gardasil — Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant Needle-free intramuscular injection, 0.5mL dose volume
  Other Names: Gardasil vial, 0.5mL
  Arms: 2: Intramuscular needle-free injection
Drug: Gardasil — Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant Needle-free intradermal injection, 0.2mL dose volume
  Other Names: Gardasil vial, 0.2mL
  Arms: 1: Intradermal needle-free injection
Device: PharmaJet Stratis® Needle-Free Injection System — 0.5mL dose injection
  Other Names: Stratis
  Arms: 2: Intramuscular needle-free injection
Device: PharmaJet Tropis® Needle-Free Injection System — 0.1mL dose injection
  Other Names: Tropis
  Arms: 1: Intradermal needle-free injection

SUMMARY:
The goal of this clinical trial is to evaluate the safety and immunogenicity of an HPV Vaccine (Gardasil) delivered by intramuscular needle-free injection and intradermal needle-free injection. The main question it aims to answer is:

* Is intramuscular and intradermal needle-free injection of Gardasil safe?
* Does intramuscular and intradermal needle-free vaccination with Gardasil illicit an immune response?

Participants will:

* Receive Gardasil by intramuscular needle-free injection, intradermal needle-free injection, or needle and syringe injection.
* Provide blood samples
* Complete physical exams
* Complete diaries

ELIGIBILITY:
Inclusion Criteria:

* Female between the age of 12 years and 13 years, inclusive. (Female 7th grade junior high school students in Indonesia)
* Clinically healthy, as established by medical history and physical examination before entering the study.
* Not pregnant at the time of vaccination.
* Able to provide informed consent and assent.
* Able to comply with the study.

Exclusion Criteria:

* Previous vaccination against HPV.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days prior to study enrollment, or planned use during the study period.
* Administration of any vaccine within 30 days prior the study enrollment, or within 30 days of study vaccination visits.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the study enrollment, or planned use during the study period.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy, or reactions likely to be exacerbated by any component of vaccine, including yeast.
* History of chronic condition(s) requiring treatment such as cancer, chronic hepatitis or kidney disease(s), diabetes, autoimmune disease. Participants with medically stable, well controlled autoimmune disease may be permitted.
* Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection.
* Received immunoglobulins and/or blood product within 90 days preceding enrollment, or planned use during the study period.
* Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., axillary temperature <37.5°C.
* Any condition that may interfere with ability to comply with trial procedures, as assessed by the Investigator.

Ages: 12 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety of fractional dose intradermal administration of Gardasil using PharmaJet Tropis® Needle-Free Injection System | Day 0 through Day 210
Immunogenicity of fractional dose intradermal administration of Gardasil using PharmaJet Tropis® Needle-Free Injection System | 28 days following each vaccination
Safety of full dose intramuscular administration of Gardasil using PharmaJet Stratis® Needle-Free Injection System | Day 0 through Day 210
Immunogenicity of full dose intramuscular administration of Gardasil using PharmaJet Stratis® Needle-Free Injection System | 28 days following each vaccination

SECONDARY OUTCOMES:
Non-inferior immunogenicity of intradermal administration of Gardasil using PharmaJet Tropis® Needle-Free Injection System compared to full dose intramuscular administration of Gardasil using needle and syringe | 28 days following each vaccination
Non-inferior immunogenicity of intramuscular administration of Gardasil using PharmaJet Stratis® Needle-Free Injection System compared to full dose intramuscular administration of Gardasil using needle and syringe | 28 days following each vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Padjadjaran, Bandung, Indonesia

IPD SHARING:
Plan to Share IPD: No